CLINICAL TRIAL: NCT05318573
Title: A Phase 2a Study With Safety Run-in to Evaluate the Safety, Tolerability, and Preliminary Efficacy of FF-10832 Monotherapy or in Combination With Pembrolizumab in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate Safety, Efficacy of FF-10832 in Combo With Pembrolizumab in Urothelial & Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujifilm Pharmaceuticals U.S.A., Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FF10832-PEM-201/KEYNOTE-B57; MK-3475-B57 (Other: Merck Sharp & Dohme Corp)
Record Dates: First submitted 2022-03-29; First posted 2022-04-08 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Advanced Urothelial Carcinoma; Advanced Non Small Cell Lung Cancer
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: FF-10832 (Gemcitabine Liposome Injection) given intravenously Day 1 of a 21-day cycle, in combination with 200 mg pembrolizumab given intravenously Day 1 of the same 21-day cycle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Safety Run-in Phase (Experimental): FF-10832 in combination therapy with pembrolizumab; FF-10832 will be dosed at 40 mg/m2 with a fixed dose of pembrolizumab (200 mg)
  Interventions: Drug: Pembrolizumab; Drug: FF-10832
- Urothelial Monotherapy - FF-10832 Expansion Phase (Experimental): FF-10832 will be dosed at 40 mg/m2
  Interventions: Drug: FF-10832
- Urothelial Combination - FF-10832 + pembrolizumab Expansion Phase (Experimental): FF-10832 in combination therapy with pembrolizumab; FF-10832 will be dosed at 40 mg/m2 with a fixed dose of pembrolizumab (200 mg)
  Interventions: Drug: Pembrolizumab; Drug: FF-10832
- NSCLC Monotherapy - FF-10832 Expansion Phase (Experimental): FF-10832 will be dosed at 40 mg/m2
  Interventions: Drug: FF-10832
- NSCLC Combination - FF-10832 + pembrolizumab Expansion Phase (Experimental): FF-10832 in combination therapy with pembrolizumab; FF-10832 will be dosed at 40 mg/m2 with a fixed dose of pembrolizumab (200 mg)
  Interventions: Drug: Pembrolizumab; Drug: FF-10832

INTERVENTIONS:
Drug: Pembrolizumab — Treatment at 200 mg pembrolizumab, administered intravenously (IV) on Day 1 of each 21-day cycle prior to infusion of FF-10832
  Other Names: KEYTRUDA®; MK-3475
  Arms: NSCLC Combination - FF-10832 + pembrolizumab Expansion Phase; Safety Run-in Phase; Urothelial Combination - FF-10832 + pembrolizumab Expansion Phase
Drug: FF-10832 — Following administration of pembrolizumab, FF-10832 Gemcitabine Liposome Injection, 40 mg/m2 administered intravenously (IV) on Day 1 of each 21-day cycle
  Other Names: Gemcitabine Liposome Injection

SUMMARY:
To confirm a recommended Phase 2 dose (RP2D) of FF-10832 (Gemcitabine Liposome Injection) given intravenously Day 1 of a 21-day cycle, in combination with 200 mg pembrolizumab given intravenously Day 1 of the same 21-day cycle, for treatment of advanced urothelial and non-small cell lung cancer

DETAILED DESCRIPTION:
This is a Phase 2a, open label clinical trial evaluating FF-10832 in combination with pembrolizumab and as monotherapy. The trial will begin with a safety run-in phase of 10 patients receiving combination therapy with pembrolizumab; FF 10832 will be dosed at 40 mg/m2 with a fixed dose of pembrolizumab (200 mg).

After confirmation of the appropriate FF-10832 dose for use with pembrolizumab, the trial will enroll up to an additional 100 patients in 2 cohorts (urothelial cancer [UC] and non-small cell lung cancer [NSCLC]) into 4 separate expansion treatment arms (approximately 25 patients in each treatment arm). The disease-defined cohorts will be patients who have progressed on PD-1/PD-L1 therapy who have UC or NSCLC.

The UC cohort will be randomized (1:1) to one of two treatment arms (monotherapy or combination therapy) and the NSCLC cohort will be randomized (1:1) to one of two treatment arms (monotherapy or combination therapy), to further establish safety and gain preliminary information on antitumor activity of FF-10832 as monotherapy or in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent is provided by patient or legally acceptable representative;
2. Age ≥ 18 years;
3. Patient populations:

   1. In the Safety Run-in, patients with histologically or cytologically confirmed advanced or metastatic solid tumors who have disease progression after treatment with standard therapies for metastatic disease that are known to confer clinical benefit, or are intolerant to treatment or refuse standard treatment will be enrolled in therapy
   2. In Expansion Phase, patient must have urothelial or NSCLC, and have failed prior anti-PD-1 or anti-PD-L1
4. Have measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology
5. Eastern Cooperative Oncology Group performance status of 0 to 1
6. Life expectancy of ≥ 3 months

Exclusion Criteria:

1. Positive urine pregnancy test within 72 hours prior to treatment
2. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks (or 5 half-lives, whichever is shorter) prior to treatment;
3. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137), AND was discontinued from that treatment due to a Grade 3 or higher immune-related adverse event;
4. Has received prior radiotherapy within 2 weeks of start of study treatment.
5. For patients with NSCLC:

   1. Patients who have received radiation therapy to the lung that is >30 Gy within 6 months of the first dose of trial treatment are excluded;
   2. Patients with mutations (e.g., EGFR mutations or ALK gene rearrangements) will be excluded unless they have been previously treated with all specific targeted therapies.
6. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention.
7. Has had an allogeneic tissue /solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Determine the incidence of Treament Emergent Adverse Events (TEAE) | 7 years
  Safety and tolerability assessed by adverse events (AEs) and serious adverse events (SAEs) and to confirm dose (RP2D) of FF-10832 given intravenously Day 1 of a 21 day cycle, in combination with 200 mg pembrolizumab, given intravenously Day 1 of the same 21-day cycle, for treatment of advanced solid tumors.
Duration of Stable Disease in Monotherapy | 7 years
  To obtain a preliminary estimate of efficacy of FF-10832 monotherapy in expansion cohorts of patients with urothelial cancer (UC) and non-small cell lung cancer (NSCLC). Duration of Stable Disease is the length of time from the start of the treatment until the criteria for progression are met
Duration of Stable Disease in Combination Therapy | 7 years
  To obtain a preliminary estimate of efficacy of the combination in expansion cohorts of patients with UC and NSCLC. Duration of Stable Disease is the length of time from the start of the treatment until the criteria for progression

SECONDARY OUTCOMES:
Determine Safety Profile of Monotherapy | 7 years
  To describe the safety profile of FF-10832 monotherapy 40 mg/m2 given intravenously Day 1 of a 21-day cycle, including treatment-emergent AEs.
  Safety assessed by adverse events (AEs) and serious adverse events (SAEs)
Determine Safety Profile of Combination Therapy | 7 years
  Describe the safety profile of the combination, including dose limiting toxicities, immune related toxicities, and other treatment emergent AEs. Safety assessed by adverse events (AEs) and serious adverse events (SAEs)
Overall Response Rate (ORR) | 7 years
  Overall Response Rate is determined by classification of solid tumors via RECIST v.1.1
Duration of Response (DOR) | 7 years
  Duration of Response is calculated from the date of first response to the date of progression or death
Progression-free survival (PFS) | 7 years
  Progression-free survival will be calculated from the date of first treatment to the date of progression or death
Overall survival (OS) | 7 years
  Overall survival will be calculated from the date of first treatment to the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Cancer and Blood Speciality Clinic, Long Beach, California
  - Sharp Memorial Hospital (Oncology Clinical Research), San Diego, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville Brown Cancer Center, Louisville, Kentucky
  - Henry Ford Cancer - Detroit (Brigitte Harris Cancer Pavilion), Detroit, Michigan
  - Washington University School of Medicine, Center for Adv Medicine, St Louis, Missouri
  - Nebraska Cancer Specialists - Legacy, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada - Southern Hills, Las Vegas, Nevada
  - Atlantic Health System / Morristown Medical Center, Morristown, New Jersey
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - TriHealth Cancer Institute; Good Samaritan Hospital, Cincinnati, Ohio
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Hospital of the Univ of Pennsylvania Perlman Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
undecided